CLINICAL TRIAL: NCT04641338
Title: Randomized, Open, Multicentre, National Superiority Clinical Trial to Assess the Combination of Fixed Dosage of Dipyrone and Codeine Compared to the Isolated Use of Components in the Control of Moderate to Severe Pain After Open Pelvic-abdominal Surgery.
Brief Title: Fixed Combination of Dipirone and Codeine Compared to the Isolated Use of Dipyrone and Codeine in Controlling Pain After Pelvic-abdominal Surgery.
Acronym: DIPICOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brazilian Clinical Research Institute (Other)
Collaborators: Brainfarma Industria Química e Farmacêutica S/A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03/2020
Record Dates: First submitted 2020-10-07; First posted 2020-11-23 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Pain, Postoperative
Keywords: Dipirone; Codeine; pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Codeine; Dipyrone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Drug: Fixed dose combination Dipyrone and Codeine
- Control group (Active Comparator)
  Interventions: Drug: Dipyrone; Drug: Codeine

INTERVENTIONS:
Drug: Fixed dose combination Dipyrone and Codeine — Fixed dose combination: dipyrone 1000 mg + codeine 30 mg every 6 hours if necessary.
  Arms: Intervention group
Drug: Dipyrone — use of 1000 mg dipyrone every 6 hours if necessary.
  Arms: Control group
Drug: Codeine — 30 mg codeine every 6 hours if necessary.
  Arms: Control group

SUMMARY:
Phase III clinical trial, multicentre of superiority, randomized, open, parallel groups, with active control and use of postoperative oral medication (multiple doses of medication).

DETAILED DESCRIPTION:
The main objective is to evaluate the effectiveness and safety of the association in relation to the isolated use of medicines.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years;
* Patients in the 1st postoperative period of open abdominal or pelvic surgery (last 24 hours) and receiving short duration analgesics or opioids in any route of administration on the previous day, being able to receive oral medication and scheduled home discharge in hours or days, with pain moderate to intense intensity (defined as VAS pain ≥ 4);
* Have signed the informed consent form.

Exclusion Criteria:

* Surgical complications to the inclusion of the participant in the research;
* Other serious comorbidities at the discretion of the investigators (such as a history of renal, hepatic, cardiac or other peptic ulcer);
* History of chronic and current use of opioids or other analgesics;
* Users of alcohol or illicit drugs;
* Use of drugs with the potential to interact with study drugs;
* Allergy, hypersensitivity or known contraindication to the use of components of the study drug;
* Psychiatric or social disorders that prevent adequate follow-up to the protocol;
* Show inability to understand and perform current pain assessments in the study;
* Women of childbearing potential, defined as all physiologically capable women of childbearing, unless they are using effective contraceptive methods while administering study medication;
* Any clinical condition that the investigator considers to generate risk to the patient or interfere with the conduct of the study;
* Participation in another clinical study in less than a year (unless participation by the principal investigator is justified).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Average of sum of the pain difference | During hospitalization (around 48 hours post surgical procedure)
  The primary endpoint of the study is the average sum of the pain difference after study medication compared to the baseline by visual analogic scale from 0 to 10 cm, where 0 = no pain, and 10 = the worst imaginable pain)

SECONDARY OUTCOMES:
Average of visual analogic scale score | During hospitalization (around 48 hours post surgical procedure)
  The average visual analogic scale score (visual analogic scale from 0 to 10 cm, where 0 = no pain and 10 = the worst imaginable pain) measured at rest and during handling in subsequent medication.
VRS (verbal scale and relief assessment pain) | During hospitalization (around 48 hours post surgical procedure)
  VRS (verbal scale and relief assessment pain) where 0 = no pain relief, 1 = mild pain relief, 2 = moderate pain relief, 3 = good pain relief and 4 = excellent pain relief)
Assessment of complete pain relief by verbal scale and relief assessment pain (VRS) | During hospitalization (around 48 hours post surgical procedure)
  Assessment of complete pain relief by verbal scale assessment of pain relief (VRS where 0 = no pain relief, 1 = mild pain relief, 2 = moderate pain relief, 3 = good pain relief, and 4 = excellent pain relief).
Need for medication of rescue | During hospitalization (around 48 hours post surgical procedure)
  Number of patients who need medication of rescue (Patients who did not experience adequate pain relief with study medication who use additional analgesics, ie, rescue medication).
Assessment of satisfaction with treatment by the participant | 14 days
  Assessment of satisfaction with treatment by the participant using a standard categorical rating scale: Patient-reported global evaluation of Eficacy (PGE) scale of 5-points where 0=poor, 1=fair, 2=good , 3=very good, and 5=excellent response to therapy).
Presence of adverse events | 14 days

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Associação Hospital de Caridade Ijuí - Núcleo de Ensino e Pesquisa, Ijuí, Rio Grande do Sul
  - Hospital Universitário São Francisco na Providência de Deus, Bragança Paulista, São Paulo
  - Santa Casa de Misericórdia de Votuporanga, Votuporanga, São Paulo